CLINICAL TRIAL: NCT00010062
Title: Study Of Post-Operative Concomitant Radio-Chemotherapy With A Continuous Infusion Of Flourouracil For Adjuvant Treatment Of Resected Pancreatic Cancer
Brief Title: Fluorouracil Plus Radiation Therapy Following Surgery in Treating Patients With Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068438; FRE-GERCOR-D98-1; EU-20022
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2007-04

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells left after surgery.

PURPOSE: Phase II trial to study the effectiveness of combining fluorouracil and radiation therapy in treating patients who have undergone surgery for pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the tolerance of adjuvant fluorouracil with concurrent radiotherapy in patients with resected pancreatic adenocarcinoma.
* Determine survival without local relapse in these patients treated with this regimen.
* Determine overall survival of these patients treated with this regimen.
* Determine the effectiveness of this adjuvant therapy in these patients.

OUTLINE: This is a multicenter study.

Patients receive high-dose radiotherapy 5 days a week for 5 weeks. Patients also receive low-dose radiotherapy 4 times a week during the last 2 weeks of the 5-week course of treatment. Patients concurrently receive fluorouracil IV continuously for 5 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed pancreatic adenocarcinoma
* Complete macroscopic resection of tumor within past 30 days
* No residual visceral or peritoneal metastasis
* Involvement of Vater's ampulla or extrahepatic bile duct allowed
* No vesicular or intrahepatic cholangiocarcinomas

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Alkaline phosphatase less than 3 times normal
* Bilirubin less than 1.5 times normal

Renal:

* Creatinine less than 1.5 times normal

Cardiovascular:

* No serious cardiac failure

Pulmonary:

* No serious respiratory failure

Other:

* No other untreatable malignant tumors
* No serious psychological, familial, social, or geographical conditions that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for pancreatic adenocarcinoma

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for pancreatic adenocarcinoma
* No prior radiotherapy in an anatomically proximal region to treatment area

Surgery:

* See Disease Characteristics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Balosso, MD, PhD, Study Chair — CHU de Grenoble - Hopital de la Tronche
Locations (30):
- France (29):
  - Clinique De Savoie, Annemasse
  - Clinique Floreal, Bagnolet
  - Clinique Tivoli, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Clinique Saint - Jean, Cagne-sur-Mer
  - Polyclinique Saint Jean, Cagnes-sur-Mer
  - Hopital Fontenoy, Chartres
  - Hopital Beaujon, Clichy
  - Hopital Louis Mourier, Colombes
  - Hopital Drevon, Dijon
  - Clinique Claude Bernard, Ermont
  - Clinique Pasteur, Évreux
  - Polyclinique Jeanne d'Arc - service de Radiotherapie Oncologie, Gien
  - CHR de Grenoble - La Tronche, Grenoble
  - Hopital Saint - Louis, La Rochelle
  - Centre Jean Bernard, Le Mans
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Hopital Laennec, Paris
  - Hopital Saint Antoine, Paris
  - CHU Pitie-Salpetriere, Paris
  - Hopital Tenon, Paris
  - Clinique Ste - Marie, Pontoise
  - Hopital Claude Gallien, Quincy-sous-Sénart
  - Polyclinique De Courlancy, Reims
  - Clinique Saint Vincent, Saint-Grégoire
  - Centre du Rouget, Sarcelles
  - C.H. Senlis, Senlis
  - Centre Medico-Chirurgical Foch, Suresnes
  - Clinique Pasteur, Toulouse
- Hopital de la Ville D'Esch-sur-Alzette, Esch-sur-Alzette, Luxembourg